CLINICAL TRIAL: NCT05238181
Title: To Validate That Pyloric or Pseudopyloric Metaplasia of the Corpus Mucosa is a Specific Pathological Feature of Autoimmune Gastritis
Brief Title: Pyloric or Pseudopyloric Metaplasia of the Corpus Mucosa in Autoimmune Gastritis
Acronym: PM_in_AIG
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Tainan Hospital, Ministry of Health and Welfare (Other)
Responsible Party: Principal Investigator, Hsiu-Chi Cheng, Professor, National Cheng-Kung University Hospital
Other Study IDs: B-ER-110-440
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Autoimmune Diseases; Helicobacter Pylori Gastritis; Anemia, Pernicious; Metaplasia; Gastritis, Atrophic
Keywords: Anemia, Pernicious; Helicobacter Pylori Gastritis; Metaplasia Intestinal; Metaplasia; Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases; Anemia, Pernicious; Metaplasia; Gastritis, Atrophic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, gastric tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The autoimmune gastritis group: Autoimmune gastritis is diagnosed if the anti-parietal cell antibody titer is positive and higher than 1:10 (ImmuGloTM COMVI mouse kidney/stomach IFA kit, Immco Diagnostics, Inc. Buffalo NY, USA).
  Interventions: Diagnostic Test: Assess pyloric or pseudopyloric metaplasia of corpus by H&E stains; Diagnostic Test: Assess pyloric or pseudopyloric metaplasia of corpus by TFF2 immunohistochemistry stains; Diagnostic Test: The assessment of corpus-predominant gastritis index (CGI), Operative Link for Gastritis Assessment (OLGA), and Operative Link on Gastric Intestinal Metaplasia assessment (OLGIM)
- The controls: The patients who are enrolled to validate pathogenesis after H. pylori infection. H. pylori infection is diagnosed by histological assessment. The matched controls are needed to be confirmed to have negative anti-parietal cell antibody.
  Interventions: Diagnostic Test: Assess pyloric or pseudopyloric metaplasia of corpus by H&E stains; Diagnostic Test: Assess pyloric or pseudopyloric metaplasia of corpus by TFF2 immunohistochemistry stains; Diagnostic Test: The assessment of corpus-predominant gastritis index (CGI), Operative Link for Gastritis Assessment (OLGA), and Operative Link on Gastric Intestinal Metaplasia assessment (OLGIM)

INTERVENTIONS:
Diagnostic Test: Assess pyloric or pseudopyloric metaplasia of corpus by H&E stains — The pathologists assess pyloric or pseudopyloric metaplasia. Pyloric or pseudopyloric metaplasia of corpus is defined as the presence of torturous deep glands in a "pseudo-pylori" pattern with focal or complete loss of parietal cells. The score of pyloric or pseudopyloric metaplasia of the corpus mucosa is ranging from 0 to 3. Score 0 is no loss of parietal cells with normal fundus gland patterns. Score 1 presents focal loss of parietal cells and scattered patterns of pyloric or pseudopyloric metaplasia with few forming pylorus-like glands. Score 2 presents focal loss of parietal cells and scattered patterns of pyloric or pseudopyloric metaplasia mixed with >= 4 pylorus-like glands. Score 3 was clusters of pylorus-like glands; the metaplasia involves > 60% of mucosa and extends to the lower third of mucosa.
  Other Names: H&E stains
Diagnostic Test: Assess pyloric or pseudopyloric metaplasia of corpus by TFF2 immunohistochemistry stains — Mouse anti-human TFF2 monoclonal antibody (R&D Systems) is used to stain gastric corpus tissues to assess the presence and degree of SPEM. The score of TFF2 staining of the corpus mucosa is ranging from 0 to 3. Score 0 is not stained. Score 1 is a "scattered" pattern of TFF staining between parietal cells; the staining is limited in the middle third of the mucosa. Score 2 is TFF2-expressing cells distributed over both the middle and lower third of the glands. Score 3 is torturous gastric oxyntic glands with a diffuse expression of TFF2 into the whole glands over both the middle and lower third of the glands of the mucosa.
  Other Names: TFF2 immunohistochemistry stains
Diagnostic Test: The assessment of corpus-predominant gastritis index (CGI), Operative Link for Gastritis Assessment (OLGA), and Operative Link on Gastric Intestinal Metaplasia assessment (OLGIM) — We take five gastric mucosal biopsies in each patient under gastroscopy, including two from the antrum (at the lesser and greater curvature, 2 cm within the pylorus, respectively), two from the corpus (at the lesser curvature of the lower corpus and the greater curvature of the middle corpus, respectively), and one from the lesser curvature of the high corpus.
  The pathologists assess the gastric pathology according to the updated Sydney system. Accordingly, the histological findings are translated into CGI, the Operative Link for Gastritis Assessment (OLGA), and the Operative Link on Gastric Intestinal Metaplasia Assessment (OLGIM) stages.
  Other Names: updated Sydney system

SUMMARY:
The study is aimed to investigate the different rates of pyloric/ pseudopyloric metaplasia or spasmolytic polypeptide-expressing metaplasia (SPEM) of corpus between autoimmune gastritis and H. pylori-infected non-ulcer dyspepsia.

DETAILED DESCRIPTION:
Autoimmune gastritis is not an uncommon disease among northern European ancestry, but its prevalence rates are unclear in other populations, including Taiwanese. A study showed that near 2% of persons more than 60 years old have undiagnosed pernicious anemia, one of the complications of autoimmune gastritis. Believed to be undiagnosed, patients are at risk of gastric malignancy and vitamin B12 deficiency-related complications until the end stage. Therefore, use of available diagnostic tools to diagnose patients with autoimmune gastritis has been important. However, autoimmune gastritis has a silent course and is not easy to be early recognized. Early recognition is important because in the late stage, vitamin B12 replacement treatment may correct pernicious anemia only but not neurologic disorders. Fundus and corpus atrophy with parietal cells loss presented 2 to 3 decades before anemia develops in autoimmune gastritis. It is no doubt that autoimmune gastritis could be diagnosed if vitamin B12 deficiency with megaloblastosis and anemia developed; however, it could be diagnosed earlier if the gastric pathological finding was noticed to be a diagnostic clue. Nevertheless, fundus and corpus atrophy is presented not only in autoimmune gastritis but also in H. pylori-related gastropathy. Therefore, we need a pathologic feature which could help physicians differentiate autoimmune gastritis from H. pylori-infected gastropathy. Here, we propose that pyloric or pseudopyloric metaplasia of corpus is distinct from H. pylori-infected gastropathy. We believe that this specific pathologic feature will be helpful to diagnose patients with autoimmune gastritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present with relevant symptoms or signs of upper gastrointestinal diseases, including, but not limited to the following: impaired gastric emptying, epigastric discomfort, postprandial bloating, early satiety, epigastric pain, acid regurgitation, dyspepsia, anemia, or vitamin B12 deficiency, or iron deficiency, are candidates to be enrolled to receive gastroscopy.

Exclusion Criteria:

* The exclusion criteria are as follows including use of aspirin, non-steroidal anti-inflammatory drugs, or cyclooxygenase-2 selective inhibitors for more than 3 months, or diagnosis with upper gastrointestinal cancer including esophagus, stomach, duodenum, mucosa-associated lymphoid tissue lymphoma, other gastric lymphoma, or pancreas.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients at the outpatient department or at the inpatient wards of National Cheng Kung University Hospital and Tainan hospital in Tainan, Taiwan, will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The pyloric or pseudopyloric metaplasia of corpus by positive TFF2 staining | 1 to 3 months after gastric biopsy
  The rates of pyloric or pseudopyloric metaplasia of corpus defined by positive TFF2 staining are compared between the two groups
The pyloric or pseudopyloric metaplasia of corpus by H&E staining | 7 days after gastric biopsy
  The rates of pyloric or pseudopyloric metaplasia of corpus defined by H&E staining are compared between the two groups.

SECONDARY OUTCOMES:
The positive corpus-predominant gastritis index | 7 days after gastric biopsy
  The rates of positive corpus-predominant gastritis index defined by updated Sydney system are compared between the two groups.
The stages of the Operative Link for Gastritis Assessment (OLGA) | 7 days after gastric biopsy
  The stages of the Operative Link for Gastritis Assessment (OLGA) defined by updated Sydney are compared between the two groups.
The stages of the Operative Link on Gastric Intestinal Metaplasia Assessment (OLGIM) | 7 days after gastric biopsy
  The stages of the Operative Link on Gastric Intestinal Metaplasia Assessment (OLGIM) defined by updated Sydney are compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Chi Cheng, MD, PhD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wada Y, Nakajima S, Kushima R, Takemura S, Mori N, Hasegawa H, Nakayama T, Mukaisho KI, Yoshida A, Umano S, Yamamoto K, Sugihara H, Murakami K. Pyloric, pseudopyloric, and spasmolytic polypeptide-expressing metaplasias in autoimmune gastritis: a case series of 22 Japanese patients. Virchows Arch. 2021 Jul;479(1):169-178. doi: 10.1007/s00428-021-03033-5. Epub 2021 Jan 30. PMID 33515301
- [Result] Tsai YC, Hsiao WH, Yang HB, Cheng HC, Chang WL, Lu CC, Sheu BS. The corpus-predominant gastritis index may serve as an early marker of Helicobacter pylori-infected patients at risk of gastric cancer. Aliment Pharmacol Ther. 2013 May;37(10):969-78. doi: 10.1111/apt.12291. Epub 2013 Apr 2. PMID 23550594
- [Result] Cheng HC, Tsai YC, Yang HB, Yeh YC, Chang WL, Kuo HY, Lu CC, Sheu BS. The corpus-predominant gastritis index can be an early and reversible marker to identify the gastric cancer risk of Helicobacter pylori-infected nonulcer dyspepsia. Helicobacter. 2017 Aug;22(4). doi: 10.1111/hel.12385. Epub 2017 Mar 22. PMID 28326664